CLINICAL TRIAL: NCT04794868
Title: Prediction and Validation of Clinical Course of Coronary Artery Disease With CT-Derived Non-Invasive Hemodynamic Phenotyping and Plaque Characterization
Brief Title: PreDiction and Validation of Clinical CoursE of Coronary Artery DiSease With CT-Derived Non-Invasive HemodYnamic Phenotyping and Plaque Characterization (DESTINY Study)
Acronym: DESTINY
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Elucid Bioimaging Inc. (Industry); Shanghai Institute of Cardiovascular Diseases (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: NCT20210308-JM
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Acute Coronary Syndrome; Ischemic Heart Disease
Keywords: acute coronary syndrome; plaque characteristics; fractional flow reserve; fractional myocardial mass
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Culprit vessel of acute coronary syndrome: Culprit vessel of acute coronary syndrome
  Interventions: Diagnostic Test: CCTA-derived high risk plaque characteristics; Diagnostic Test: CFD-derived hemodynamic parameters
- Non-culprit vessel of acute coronary syndrome: Non-culprit vessel of acute coronary syndrome
  Interventions: Diagnostic Test: CCTA-derived high risk plaque characteristics; Diagnostic Test: CFD-derived hemodynamic parameters

INTERVENTIONS:
Diagnostic Test: CCTA-derived high risk plaque characteristics — Presence of CCTA-derived high risk plaque characteristics
Diagnostic Test: CFD-derived hemodynamic parameters — CFD-derived hemodynamic parameters

SUMMARY:
Acute coronary syndrome (ACS) and sudden cardiac death can be the first manifestation of coronary artery disease and are the leading cause of death in the majority of the world's population. The main pathophysiology of ACS is well-known and fibrous cap thickness, presence of a lipid core, and the degree of inflammation have been proposed as the key determinants of plaque vulnerability. Previous studies using virtual histology intravascular ultrasound or optical coherence tomography showed that clinical application of this concept improved risk prediction of ACS. However, these approaches have not been widely adopted in daily practice due to relatively low positive predictive values, low prevalence of high-risk plaques and the invasive nature of diagnostic modalities.

Non-invasive imaging studies with coronary computed tomography angiography (CCTA) also showed the clinical value of CCTA-derived high risk plaque characteristics (HRPC). In addition, the recent progress in CCTA and computational fluid dynamics (CFD) technologies enables simultaneous assessment of anatomical lesion severity, presence of HRPC and quantification of hemodynamic forces acting on plaques in patient-specific geometric models. As plaque rupture is a complicated biomechanical process influenced by the structure and constituents of the plaque as well as the external mechanical and hemodynamic forces acting on the plaque, a comprehensive evaluation of lesion geometry, plaque characteristics and hemodynamic parameters may enhance the identification of high-risk plaque and the prediction of ACS risk.

In this regard, the current study is designed to evaluate prognostic implications of comprehensive non-invasive hemodynamic assessment using CCTA and CFD in the identification of high risk plaques that caused subsequent ACS.

DETAILED DESCRIPTION:
The study population was collected from Samsung Medical Center. Target population is patients who suffered a clearly documented ACS (acute myocardial infarction [MI] or unstable angina with objective evidence of plaque rupture) or those who underwent significant lesion progression in angiography and treated by percutaneous coronary intervention (PCI) and had undergone CCTA from 6 months to 3 years prior to the coronary events.

CCTA images were screened for plaque characteristics and CFD analysis at core laboratories in Elucid Bioimaging, Inc, MA, USA and Shanghai Institute of Cardiovascular Diseases, Shanghai, China, respectively. Lesions with diameter stenosis (DS) > 30% based on CCTA evaluation were included analysis. The presence of conventional CCTA-HRPC (minimum lumen area<<4 mm2, plaque burden≥70%, low-attenuation plaque, positive remodeling, napkin-ring sign, and spotty calcification) and parameters from tissue characterization using VascuCAP software will be assessed in each lesion by an independent observer blinded to the clinical data and CFD results. The hemodynamic parameters from CFD will include 1) per-vessel FFR derived from CCTA (FFRCT); 2) change in FFRCT across the lesion (△FFRCT); 3) FFRCT pullback pressure gradient (PPG) index (FFRCT-PPG index); 4) Fractional myocardial mass (FMM) of the target stenosis.

Using the occurrence of ACS or PCI for the progressed lesion as clinical endpoint, prognostic implications of CCTA-derived HRPC or hemodynamic parameters will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who presented with ACS and underwent invasive coronary angiography with identifiable culprit lesion
2. Patients who presented with stable ischemic heart disease and underwent invasive coronary angiography for the significant epicardial coronary stenosis
3. The patients who underwent coronary CT angiography, regardless of the reason (for example, routine healthcare check-up, or evaluation for stable angina or atypical chest pain) prior to the acute event.
4. Time limit of CCTA: 6 months ~ 3 years prior to the event.
5. Definition of ACS:

   * The patients with acute myocardial infarction should meet one of the following criteria;

     * Cardiac enzyme elevation "and"
     * Identified culprit lesion confirmed by invasive coronary angiography, IVUS, or OCT
   * The patients with unstable angina should be accompanied by the evidence of plaque rupture confirmed with invasive coronary angiography, IVUS, or OCT

Exclusion Criteria:

Exclusion criteria for Patient enrollment

* Patients with acute coronary syndrome without clear evidence of culprit lesion
* Patients with stents in two or more vessel territories prior to CCTA
* Poor quality of CCTA which is unsuitable for plaque and CFD analysis
* Patients with ACS culprit lesion in a stented vessel
* Patients with previous history of coronary artery bypass graft surgery
* Secondary myocardial infarction due to other general medical conditions, such as sepsis, arrhythmia, bleeding, etc.
* Poor quality CCTA images unsuitable for CFD analysis
* No available unprocessed CCTA data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population was collected from Samsung Medical Center. Target population is patients who suffered a clearly documented ACS (acute myocardial infarction [MI] or unstable angina with objective evidence of plaque rupture) or those who underwent significant lesion progression in angiography and treated by percutaneous coronary intervention (PCI) and had undergone CCTA from 6 months to 3 years prior to the coronary events.
Sampling Method: Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Acute myocardial infarction | 3 years after index CCTA
  Target vessel-related acute myocardial infarction
Revascularization | 3 years after index CCTA
  Target vessel-related revsacularization

SECONDARY OUTCOMES:
Target vessel failure | 3 years after index CCTA
  A composite of Cardiac death, Target vessel-related acute myocardial infarction, Target vessel-related revsacularization
All-cause death | 3 years after index CCTA
  All-cause death
Cardiac death | 3 years after index CCTA
  Death due to cardiac cause
Major adverse cardiac and cerebral events | 3 years after index CCTA
  A composite of All-cause death, Target vessel-related acute myocardial infarction, Target vessel-related revsacularization, Cerebrovascular accident

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (2):
- Shanghai Institute of Cardiovascular Diseases, Shanghai, China
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Anatomized patient data can be shared upon reasonable request after decision by principal investigator

REFERENCES:
- [Derived] Hong D, Dai N, Lee SH, Shin D, Choi KH, Kim SM, Kim HK, Jeon KH, Ha SJ, Lee KY, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Choe YH, Gwon HC, Ge J, Lee JM. Fractional Flow Reserve and Fractional Flow Reserve Gradient From CCTA for Predicting Future Coronary Events. JACC Asia. 2024 Aug 27;4(10):735-747. doi: 10.1016/j.jacasi.2024.06.007. eCollection 2024 Oct. PMID 39553907
- [Derived] Lee SH, Hong D, Dai N, Shin D, Choi KH, Kim SM, Kim HK, Jeon KH, Ha SJ, Lee KY, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Choe YH, Gwon HC, Ge J, Lee JM. Anatomic and Hemodynamic Plaque Characteristics for Subsequent Coronary Events. Front Cardiovasc Med. 2022 May 23;9:871450. doi: 10.3389/fcvm.2022.871450. eCollection 2022. PMID 35677691